CLINICAL TRIAL: NCT03125538
Title: Therapeutic Effects of Motor Imagery Practice Following Lower-limb Amputation
Brief Title: Motor Imagery Practice on Amputees (MIPA)
Acronym: MIPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratoire Interuniversitaire de Biologie de la Motricité (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: Libm
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Rehabilitation
Keywords: Motor Imagery; Amputation; Functional rehabilitation; Locomotion; Phantom-limb pain
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Intervention Model Description: To avoid group contamination, a first group of 10 control participants will be completed. Then, an experimental group of 10 patients will be assessed. In order to complete a 40 persons cohort, this will be repeated one time (other 10 control then 10 experimental participants).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants sign an informed written consent but are not aware of the expectations of the study. Assessments will be performed by a PhD student who does not know neither to which group each participants belongs, nor the expectations of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Imagery (Experimental): Participants from the experimental group will perform MIP concomitantly with usual physical rehabilitation program.
  Interventions: Other: Motor Imagery
- Control task (Active Comparator): Concomitantly with usual physical rehabilitation program, participants from the control group will perform a cognitive task that has no impact on motor rehabilitation (word scramble game).
  Interventions: Other: Control Task

INTERVENTIONS:
Other: Motor Imagery — Together with physical rehabilitation performed with physiotherapists, participants from the experimental group will mentally rehearse 3 different locomotor exercises that they already physically performed beforehand.
  Exercise 1: 10m Walk
  Exercise 2: Timed Up and Go test (rise up from a chair, walk 3 meters, turn around, come back to the chair, turn around and sit down)
  Exercise 3: Stairs climbing test (climb up 4 stairs, turn around, climb down the for stairs)
  Two min of MIP will be scheduled 5 times/day, during rest periods, so that patients complete 10min of MIP per day.
  Arms: Motor Imagery
Other: Control Task — Together with physical rehabilitation performed with physiotherapists, participants from the control group will spend equivalent time focusing on a cognitive task without impact on motor rehabilitation ((word scramble game).
  Two min of this cognitive task will be scheduled 5 times/day, during rest periods, so that patients complete 10min of control task per day.
  Arms: Control task

SUMMARY:
Motor imagery practice (MIP), which is the repeated internal representation of a movement without engaging its physical execution and which shares a neurofunctional equivalence with physical practice, has been show to contribute to promote motor recovery and pain alleviation. Despite the extensive body of evidence concerning MIP therapeutic effects, the impact of mental training during lower-limb amputees' rehabilitation process remains to be investigated. This study was designed to assess MIP effects on the relearning of walking and the frequency and intensity of phantom-limb pain among acute lower-limb amputees. Data should contribute to scale up the tools made available to therapists and extend the scope of MIP application. Moreover, results may contribute to directly provide patients recovering from a lower-limb amputation with a cost-effective and adaptable technique that could considerably improve their quality of life.

DETAILED DESCRIPTION:
Arms:

Arm label: Experimental

Arm type: Experimental

Arm description: Participants from the experimental group will perform MIP concomitantly with usual physical rehabilitation program.

Intervention type: Other

Intervention name: Motor Imagery Practice of locomotor tasks

Intervention Description: Together with physical rehabilitation performed with physiotherapists, participants from the experimental group will mentally rehearse 3 different locomotor exercises that they already physically performed beforehand.

Exercise 1: 10m Walk

Exercise 2: Timed Up and Go test (rise up from a chair, walk 3 meters, turn around, come back to the chair, turn around and sit down)

Exercise 3: Stairs climbing test (climb up 4 stairs, turn around, climb down the for stairs)

Two min of MIP will be scheduled 5 times/day, during rest periods, so that patients complete 10min of MIP per day.

Locomotor capacities and phantom-limb pain intensity will be assessed at 5 different moments of the functional rehabilitation:

Evaluation 1: first day of functional rehabilitation Evaluation 2: right after prosthesis fitting and when patients are able to walk with it during 10min Evaluation 3: three weeks after the second evaluation (to have temporally equivalent data for all patients) Evaluation 4: one week before leaving the rehabilitation center (to have functionally equivalent data for all patients) Evaluation 5: six weeks after patients left the center, for follow-up assessment

Arm label: Control

Arm type: Active comparator

Arm description: Concomitantly with usual physical rehabilitation program, participants from the control group will perform a cognitive task that has no impact on motor rehabilitation (word scramble game).

Intervention type: Other

Intervention name: Control cognitive task

Intervention Description: Together with physical rehabilitation performed with physiotherapists, participants from the control group will spend equivalent time focusing on a cognitive task without impact on motor rehabilitation.

Two min of this cognitive task will be scheduled 5 times/day, during rest periods, so that patients complete 10min of control task per day.

As for patients of the experimental group, locomotor capacities and phantom-limb pain intensity of participants from the control group will be assessed at 5 different moments of the functional rehabilitation:

Evaluation 1: first day of functional rehabilitation Evaluation 2: right after prosthesis fitting and when patients are able to walk with it during 10min Evaluation 3: three weeks after the second evaluation (to have temporally equivalent data for all patients) Evaluation 4: one week before leaving the rehabilitation center (to have functionally equivalent data for all patients) Evaluation 5: six weeks after patients left the center, for follow-up assessment

ELIGIBILITY:
Inclusion Criteria:

* Suffering from acute transtibial or transfemoral lower-limb amputation
* Having signed informed consent for an clinical study
* Having a score above 24/30 at the Mini Mental Status Examination

Exclusion Criteria:

* Persons under any administrative/judicial measure
* Participants refusing to be informed of the results of the experiment
* Persons with other motor impairments
* Persons with neurologic and/or psychiatric disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02-25 (Actual); Primary Completion 2017-10-30 (Estimated); Study Completion 2017-10-30 (Estimated)

PRIMARY OUTCOMES:
MIP effects on simple walking | From first day of functional rehabilitation until patients leave the center (approximately from 6 to 10 weeks depending on their ability to recover enough functional autonomy)
  Duration required to perform a 10m walk will be assessed at 1) patients first day of functional rehabilitation, 2) right after prosthesis fitting and when they are able to walk with it during 10min, 3) three weeks after the second evaluation (to have temporally equivalent data for all the patients), 4) one week before leaving the rehabilitation center (to have functionally equivalent data for all patients), and 5) six weeks after patients left the center, for follow-up assessment.
MIP effects on the Timed Up and Go test (complex walking task involving turning, and raise and sit movements) | From first day of functional rehabilitation until patients leave the center (approximately from 6 to 10 weeks depending on their ability to recover enough functional autonomy)
  Duration required to perform the test Timed Up and Go will be assessed at 1) patients first day of functional rehabilitation, 2) right after prosthesis fitting and when they are able to walk with it during 10min, 3) three weeks after the second evaluation (to have temporally equivalent data for all the patients), 4) one week before leaving the rehabilitation center (to have functionally equivalent data for all patients), and 5) six weeks after patients left the center, for follow-up assessment.
MIP effects on a climbing locomotor task | From first day of functional rehabilitation until patients leave the center (approximately from 6 to 10 weeks depending on their ability to recover enough functional autonomy)
  Duration required to perform 4 stairs climbing test (up and down) will be assessed at 1) patients first day of functional rehabilitation, 2) right after prosthesis fitting and when they are able to walk with it during 10min, 3) three weeks after the second evaluation (to have temporally equivalent data for all the patients), 4) one week before leaving the rehabilitation center (to have functionally equivalent data for all patients), and 5) six weeks after patients left the center, for follow-up assessment.

SECONDARY OUTCOMES:
Phantom-limb pain | From first day of functional rehabilitation until patients leave the center (approximately from 6 to 10 weeks depending on their ability to recover enough functional autonomy)
  Patients will rate from 0 (no pain at all) to 100 (the worst pain possible), the intensity of the phantom-limb pain they experienced during the last 24h. Assessment will be performed during the 5 evaluations, as described for the primary outcome measure.
Motor imagery time | From first day of functional rehabilitation until patients leave the center (approximately from 6 to 10 weeks depending on their ability to recover enough functional autonomy)
  The time required to imagine the three locomotor tasks (walking, Timed Up and Go and stairs climbing tests) and a simple movement (hip abduction) will be recorded. Assessment will be performed during the 5 evaluations, as described for the primary outcome measure.
Motor imagery vividness | From first day of functional rehabilitation until patients leave the center (approximately from 6 to 10 weeks depending on their ability to recover enough functional autonomy)
  The capacity of patients to perform vivid MI (clear images and intense kinesthetic sensations while imaging) will be measured with the Kinesthetic and Visual Motor Imagery Questionnaire. Assessment will be performed during the 5 evaluations, as described for the primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Aymeric Guillot, Professor, Principal Investigator — Laboratoire Interuniversitaire de Biologie de la Motricité
Locations (1):
- Centre Médico-Chirirgical de Réadaptation des Massues, Lyon, Rhône, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saruco E, Saimpont A, Di Rienzo F, De Witte B, Laroyenne I, Mateo F, Lapenderie M, Solard SG, Perretant I, Frenot C, Jackson PL, Guillot A. Towards efficient motor imagery interventions after lower-limb amputation. J Neuroeng Rehabil. 2024 Apr 15;21(1):55. doi: 10.1186/s12984-024-01348-3. PMID 38622634